CLINICAL TRIAL: NCT00704704
Title: A Phase 2, Single Arm Study to Determine the Safety and Efficacy of Azacitidine, and Thalidomide in Higher Risk Myelodysplastic Syndrome
Brief Title: Safety and Efficacy of Azacitidine, and Thalidomide in Higher Risk MDS (Myelodysplastic Syndrome)
Acronym: IMDS001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-08-MM-TLV-0069-08-CTIL
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: high risk MDS; IPSS; 5-AZA-Cytidine; Thalidomide; response rate; cytogenetic response; QOL questionaries; INT-2 or High risk MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 5-aza-cytidine and Thalidomide — 5-AZA-Cytidine 75mg/m2 5 days a month. 12 months. Thalidomide 50mg orally daily for 6 months.
  Other Names: vidaza

SUMMARY:
Study Objectives The aim of the study is to evaluate the safety and efficacy of the combination of 5-Aza-Cytidine + Thalidomide on the course of hrMDS patients.

Primary end point:

• To evaluate the overall response rate (CR+PR) of the combination of 5-Aza-Cytidine + Thalidomide in hrMDS patients (INT-2 and High risk as defined by IPSS).

Secondary end points:

* To evaluate the safety of the combination of Thalidomide+5-Aza-Cytidine in high risk MDS patients.
* Hematological improvement rate.
* Cytogenetic response.
* Progression free survival (PFS).
* Quality of life assessment (FACT: MDS and peripheral neuropathy QOL Questionnaires).

Study design:

This is a multicenter, phase II, single arm study designed to evaluate the safety and efficacy of the combination of Thalidomide+5-Aza-Cytidine in high risk MDS patients (INT-2 and High risk defined by IPSS) who are older than 18 years of age. Potential study subjects will sign an informed consent prior to undergoing any study related procedure. Number of patients to be enrolled 50.

Treatment plan: 5-aza-cytidine (75 mg m2/d) will be injected subcutaneously in 5-day cycle every 28 days, for a total of 12 cycles.

Thalidomide will be given at the dose of 50 mg/d, from day 1 until for 6 months together with 5-aza-cytidine .

Treatment period includes 5-aza-cytidine (75 mg m2/d) will be injected subcutaneously in 5-day cycle every 28 days. Total number of 12 cycles or until progression or toxicity. Cycle delay of maximum 2 weeks in case of hematological toxicity grade 3-4 at investigator discretion.

Duration of the follow up period is 6 months. Duration of study The duration of the treatment period is approximately 12 months. This time is required to complete the treatment, and to determine the safety profile and the response rate. The duration of the Follow period will be approximately a half year. The occurrence of PD will determine the duration of progression-free survival of each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patient is older than 18 years at the time of signing the informed consent.
* Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable double method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Female of childbearing potential must have a negative serum β-human chorionic gonadotropin ( beta sub unit-HCG) pregnancy test both 24 hours prior to beginning of therapy and then at 4 weeks intervals in women with regular menstrual cycles or every 2 weeks in women with irregular menstrual cycles during study treatment for subjects of childbearing potential.
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of thalidomide therapy.
* Patient was diagnosed with myelodysplastic syndrome INT-2 or High risk according IPSS score .Bone marrow aspiration examination including cytogenetics performed up to 12 months before patient signing informed consent.
* Patient has a Performance Status 0-2 (WHO).
* Patient has a life-expectancy > 6 months
* Patient has not known active infectious hepatitis type B or C, or HIV infection.
* Patient is epopoietin resistant. Erythropoietin should be discontinued 28 days before starting treatment period.
* Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1):

  * Platelet count ≥ 25 x 109/L without transfusion support within 7 days before the test.
  * Absolute neutrophil count (ANC) ≥ 0.5 x 109/L without the use of growth factors.
  * Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal (ULN).
  * Alanine transaminase (ALT): ≤ 2.5 x the ULN.
  * Total bilirubin: ≤ 1.5 x the ULN.
  * Serum creatinine< 2 X the ULN.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
overall response rate measured by complete blood counts and bone marrow examinations | at study entry. after 6 months and after one year
overall response rate | 6 and 12 months

SECONDARY OUTCOMES:
*safety *hematological improvement *cytogenetic response *progression free survival * Quality of life assessment (FACT: MDS and peripheral neuropathy QOL Questionnaires). | at entry , 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hematolpgical department Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] 1. Greenberg PL. Risk factors and their relationship to prognosis in myelodysplastic syndromes. Leuk Res. 1998;22 Suppl 1:S3-6. 2. Sanz GF, Sanz MA, Greenberg PL. Prognostic factors and scoring systems in myelodysplastic syndromes. Haematologica. 1998;83:358-368. 3. Hellstrom-Lindberg E, Ahlgren T, Beguin Y, et al. Treatment of anemia in myelodysplastic syndromes with granulocyte colony-stimulating factor plus erythropoietin: results from a randomized phase II study and long-term follow-up of 71 patients. Blood. 1998;92:68-75. 4. Silverman LR, Demakos EP, Peterson BL, et al. Randomized controlled trial of azacitidine in patients with the myelodysplastic syndrome: a study of the cancer and leukemia group B. J Clin Oncol. 2002;20:2429-2440. 5. Silverman LR, McKenzie DR, Peterson BL, et al. Further analysis of trials with azacitidine in patients with myelodysplastic syndrome: studies 8421, 8921, and 9221 by the Cancer and Leukemia Group B. J Clin Oncol. 2006;24:3895-3903. 6.